CLINICAL TRIAL: NCT07403617
Title: Ventilation-Perfusion Discrepancy Index Versus Conventional Anatomic-Physiologic Assessment for Target Lung Lobe Selection in Endobronchial Valve Placement: A Multicenter, Randomised Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Principal Investigator, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SELECTION-I
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Emphysema
Keywords: Endobronchial Lung Volume Reduction; Ventilation-Perfusion Discrepancy Index; Emphysema; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VQDI-assisted target lung lobe selection strategy (Experimental): Target lobe selection is based on the lobe with the lowest VQDI among all lobes with an absence of collateral ventilation (Chartis-negative), indicating the most severe ventilation-perfusion mismatch.
  Interventions: Procedure: VQDI-assisted target lung lobe selection strategy
- Conventional target lung lobe selection strategy (Placebo Comparator): Target lobe selection is based on the lobe with the highest CT destruction score among all lobes with an absence of collateral ventilation (Chartis-negative), indicating the most severe anatomical destruction.
  Interventions: Procedure: Conventional target lung lobe selection strategy

INTERVENTIONS:
Procedure: VQDI-assisted target lung lobe selection strategy — Participants in this arm undergo endobronchial valve (EBV) placement in a target lobe selected specifically based on functional imaging. Among all lobes confirmed to have no collateral ventilation (assessed by the Chartis system), the lobe with the lowest Ventilation-Perfusion Discrepancy Index (VQDI) - indicating the most severe mismatch between air flow and blood flow - is chosen for treatment. All other procedural aspects, screening assessments, and follow-up are identical to the comparator arm.
  Arms: VQDI-assisted target lung lobe selection strategy
Procedure: Conventional target lung lobe selection strategy — Participants in this arm undergo endobronchial valve (EBV) placement in a target lobe selected based on standard anatomical criteria. Among all lobes confirmed to have no collateral ventilation (assessed by the Chartis system), the lobe with the highest CT destruction score - indicating the most severe anatomical emphysema - is chosen for treatment. This reflects current standard-of-care practice. All other procedural aspects, screening assessments, and follow-up are identical to the experimental arm.
  Arms: Conventional target lung lobe selection strategy

SUMMARY:
The goal of this clinical trial is to learn if a Ventilation-Perfusion Discrepancy Index (VQDI)-guided strategy for selecting the target lung lobe can improve outcomes compared to the standard strategy in patients with severe emphysema undergoing bronchoscopic lung volume reduction with endobronchial valves (EBVs).

The main question it aims to answer is:

· Does selecting the target lobe based on the lowest VQDI (indicating the worst functional mismatch) lead to a higher rate of successful treatment response at 6 months compared to selecting the lobe based on the worst destruction on CT scan?

If there is a comparison group: Researchers will compare the VQDI-guided selection group to the conventional CT/Chartis-guided selection group to see which strategy results in more patients achieving significant improvement in both lung function and reduction in the size of the treated lobe.

Participants will:

* Undergo standard clinical assessments (lung function tests, CT scan, exercise test) and an additional V/Q SPECT/CT scan to calculate the VQDI.
* Have their collateral ventilation status checked using the Chartis system during bronchoscopy.
* Be randomly assigned to one of the two target lobe selection strategies.
* Receive EBV placement in the selected lobe.
* Attend follow-up visits at 1, 3, 6, and 12 months after the procedure for check-ups, repeated lung function tests, questionnaires, and CT scans to assess their response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological evidence of emphysema
* Nonsmoking for 4 months prior to screening interview
* BMI less than 35 kg/m2
* Stable on current medication regimen
* Forced expiratory volume in one second (FEV1) between 15% and 45% of predicted value
* Residual Volume less than 175% predicted (determined by body plethysmography)
* Little or no collateral ventilation (CV-) as determined using the Chartis System

Exclusion Criteria:

* Had two or more hospitalizations over the last year for a COPD exacerbation
* Had two or more hospitalizations over the last year for pneumonia
* Had a prior lung transplant, lung volume reduction surgery, bullectomy or lobectomy
* Had a heart attack or congestive heart failure within the last 6 months
* Have heart arrhythmia
* Is alpha-1 antitrypsin deficient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Ventilation-Perfusion Discrepancy Index (VQDI) | 6 month
  The absolute change in the target lobe's VQDI from baseline to 6 months post-procedure.

SECONDARY OUTCOMES:
St. George's Respiratory Questionnaire (SGRQ) | 1 year
  Difference between study arms in 'absolute change from baseline' for SGRQ score at 1 year (value at 1 year minus value at baseline). The St. George's Respiratory Questionnaire measures health status (quality of life) in patients with diseases of airways obstruction. The questionnaire comprises of two parts: Part I: Symptoms (frequency & severity) Part II: Activities that cause or are limited by breathlessness; Impacts (social functioning, psychological disturbances resulting from airways disease) A Total score is calculated which summarizes the impact of the disease on overall health status. Scores range from 0 to 100, with higher scores indicating more limitations.
FEV1 Post-bronchodilator Absolute Change | 1 year
  Difference between study arms in absolute change from baseline for post-bronchodilator FEV1 score at 1 year (value at 1 year minus value at baseline).
6-minute Walk Distance | 1 year
  Difference between study arms in 'absolute and percentage change from baseline' for 6MWD at 1 year (value at 1 year minus value at baseline).

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No